CLINICAL TRIAL: NCT01973062
Title: Phase II Study of Radioimmunotherapy With Zevalin (Ibritumomab Tiuxetan) Therapy for Patients With Refractory or Relapsed Primary Central Nervous System Lymphoma (PCNSL)
Brief Title: Yttrium Y 90 Ibritumomab Tiuxetan and Rituximab in Primary Central Nervous System Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding Unavailable
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE4413; NCI-2013-01993 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Primary Central Nervous System Non-Hodgkin Lymphoma
MeSH Terms: interventions — Rituximab; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rituximab and yttrium Y 90 ibritumomab tiuxetan (Experimental): Patients receive rituximab IV on day 1. Within 7 to 9 days, patients receive rituximab IV and yttrium Y 90 ibritumomab tiuxetan IV in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Radiation: yttrium Y 90 ibritumomab tiuxetan

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Radiation: yttrium Y 90 ibritumomab tiuxetan — Given IV
  Other Names: 90Y ibritumomab tiuxetan; IDEC Y2B8; Y90 Zevalin; Y90-labeled ibritumomab tiuxetan

SUMMARY:
This phase II trial studies how well yttrium Y 90 ibritumomab tiuxetan and rituximab work in treating patients with recurrent or refractory primary central nervous system non-Hodgkin lymphoma. Radiolabeled monoclonal antibodies, such as yttrium 90 ibritumomab tiuxetan, can find cancer cells and carry cancer-killing substances to them without harming normal cells. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving yttrium Y 90 ibritumomab tiuxetan with rituximab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the radiographic response proportion in patients with refractory or recurrent primary central nervous system lymphoma (PCNSL) to ibritumomab tiuxetan (yttrium Y 90 ibritumomab tiuxetan) when given as an intravenous infusion.

SECONDARY OBJECTIVES:

I. Determine the progression free survival of patients treated with ibritumomab tiuxetan when given as an intravenous infusion.

II. Determine the overall survival of patients treated with ibritumomab tiuxetan when given as an intravenous infusion.

III. Establish the toxicity profile of ibritumomab tiuxetan in this patient population.

IV. Use positron emission tomography (PET)/magnetic resonance imaging (MRI) to map the distribution of Y-90 ibritumomab tiuxetan, and calculate the Gy delivered based on the activity found within tumor.

OUTLINE:

Patients receive rituximab intravenously (IV) on day 1. Within 7 to 9 days, patients receive rituximab IV and yttrium Y 90 ibritumomab tiuxetan IV in the absence of disease progression or unacceptable toxicity. Distribution and dose absorbed dose will be assessed on day 11. Quality of life will be assessed at screening, at day 1, 36, 92, and at each follow-up visit.

After completion of study treatment, patients are followed every 3-6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological diagnosis of recurrent or refractory primary central nervous system (CNS) lymphoma with at least 1 measurable gadolinium enhancing lesion on brain MRI scans
* Karnofsky performance status (KPS) >= 60
* Patients could not have had more than 3 prior therapy regimens for the treatment of PCNSL
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin (Hgb) > 10 g/dL
* Serum total bilirubin =< 1.5 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) =< 3.0 x ULN
* Aspartate aminotransferase (AST) =< 3.0 x ULN
* Serum creatinine =< 1.5 x ULN
* Minimum interval since completion of radiation treatment is 12 weeks
* Minimum interval since last drug therapy:

  * 3 weeks since the completion of non-cytotoxic agents
  * 4 weeks since the completion of a non-nitrosourea-containing regimen
  * 6 weeks since the completion of a nitrosourea-containing regimen
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients are not on corticosteroids or on stable doses (less than 6 mg daily of dexamethasone) for more than 1 week before baseline imaging
* Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception
* Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix and breast, adequately treated stage I or II cancer from which the patient is in complete remission; patients with other prior malignancies must be disease-free for >= three years

Exclusion Criteria:

* Pregnant or breast-feeding women
* Patients unwilling or unable to comply with the protocol
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g. active infection, uncontrolled diabetes, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, or psychiatric illness, etc.) that could cause unacceptable safety risks or compromise compliance with the protocol
* Known diagnosis of human immunodeficiency virus (HIV) infection; prior radioimmunotherapy, prior myeloablative therapy with autologous bone marrow transplantation or peripheral stem cell rescue, and prior external beam radiation therapy to more than 25% of active bone marrow
* Patients who have received filgrastim (G-CSF) or sargramostim (GM-CSF) within 2 weeks before treatment or major surgery within the prior 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manmeet Ahluwalia, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Response Assessed by MRI or FDG-PET/MRI
Description: Number of patients with at least a 50% reduction in tumor size on a MRI scan with stable or decreasing dose of corticosteroids
Time Frame: Up to 2 years
Population: Only one patient registered. No patient data analyzed
Arm/Group | Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression Free Survival
Description: The number of patients without an unequivocal increase in tumor size or the appearance of new lesions by MRI
Time Frame: Up to 2 years
Population: Only one patient registered. No patient data analyzed
Arm/Group | Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: The number of patients alive up to two years after treatment
Time Frame: Up to 2 years
Population: Only one patient registered. No patient data analyzed
Arm/Group | Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan
Number analyzed (Participants) | 0

4. Secondary Outcome: Establish the Toxicity Profile of Ibritumomab Tiuxetan in This Patient Population.
Description: Number of patients with toxicities related to the study drug
Time Frame: Up to 30 days following the last dose of study treatment
Population: Only one patient registered. No patient data analyzed
Arm/Group | Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan
Number analyzed (Participants) | 0

5. Secondary Outcome: Dosimetry Calculations of Yttrium Y 90 Ibritumomab Tiuxetan Assessed by PET/MRI
Description: Number of Gy delivered to each tumor as calculated using the MIRD dosimetry formula on PET data
Time Frame: At day 11
Population: Only one patient registered. No patient data analyzed
Arm/Group | Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes